CLINICAL TRIAL: NCT02766153
Title: Exploring the Mechanisms of Resistance of Stem Cells Myeloproliferative Opposite of Tyrosine Kinase Inhibitors in 3d Model Niche Endosteal
Status: Terminated | Type: Observational
Why Stopped: the investigator has left the hospital
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-02
Record Dates: First submitted 2016-04-20; First posted 2016-05-09 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2018-06

CONDITIONS: Myeloproliferative Disorders
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients
- healthy volunteers: intrafamily marrow donors

SUMMARY:
Myeloproliferative disorders (MPD) include chronic myeloid leukemia (CML) (Ph +) and essential thrombocythemia (ET), the polycythemia vera (PV), myelofibrosis (MF) called SMP Ph. CML is the ultimate model of carcinogenesis. SMP is a characterized by a malignant monoclonal proliferation of a pluripotent hematopoietic progenitor determined by the presence of a balanced translocation between chromosomes 9 and 22 (Ph chromosome) which leads to major changes of a large number of cell functions. Investigators now believe that within the bone marrow exist two types of "hematopoietic niches' niche osteoblastic / endosteal and vascular niche, controlling the maintenance and differentiation of hematopoietic stem cell pool. The endosteal niche, is a hypoxic region near the endosteal trabecular, which provides protection to deeply dormant stem cells. Data from the literature suggest that in the SMP, especially CML, the interaction of malignant stem cells with the microenvironment niche Endosteal could favor their survival and resistance to treatment. The therapeutic management of CML was upset by the use of tyrosine kinase inhibitors (TKIs). However, despite these advances, even in situations of undetectable residual disease, it has been observed relapses of the disease stopped TKI leaving suggest that there is a resistance of leukemic stem cell to TKI.

Work in the group Bipoa "Bio Engineering and Pathophysiology Osteo-Articular" helped develop a 3D model of ex vivo bone formation, which can mimic the endosteal niche. the goal is to apply this model to the SMP of hematopoiesis by referring to normal hematopoiesis. it will be tested the hypothesis that the endosteal ex vivo recess of the 3D modeling allows to highlight a special interaction can promote the persistence of the leukemia stem cell despite the use of effective therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LLC (chronic myeloid leukemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients selected for this study, which will continue over a period of five years, corresponding to all newly diagnosed patients or SMP during TKI treatment in the clinical hematology department of Nice University Hospital and associated centers. The recruitment of three years should be 200 patients. Healthy donors are intra-family donor marrow taken to operating room under general anesthesia as part of their marrow donation. These healthy donors have also already signed a consent for their donation, including research referred to levies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Characteristics of cell CD34 + tumor from patients with SMP | 5 years
  Establishment of a stem cell CD34 + tumor bank from patients with SMP

SECONDARY OUTCOMES:
Characteristics of the variation of TKI on CD4+ stem cells | 5 years
  Compare in vitro, in traditional culture or in a 3D environment mimicking endosteal niche, the effect of first and second generation TKIs on CD34 + stem cells made from patients with SMP or healthy volunteer donors

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France